CLINICAL TRIAL: NCT04797390
Title: A Randomized Trial of an Advanced Pneumatic Compression Device vs. Usual Care for Head and Neck Lymphedema
Brief Title: A Study Evaluating an Advanced Pneumatic Compression Device Versus Usual Care for Treatment of Head and Neck Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tactile Medical (Industry)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8030
Record Dates: First submitted 2021-03-05; First posted 2021-03-15 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2024-05

CONDITIONS: Lymphedema; Lymphedema of Face; Lymphedema, Secondary; Lymphedema Due to Radiation; Lymphedema; Surgical
Keywords: Head and Neck Lymphedema
MeSH Terms: conditions — Lymphedema; Neoplasm Metastasis | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Advanced Pneumatic Compression Device (APCD) (Active Comparator): Daily self-administered treatment with the Flexitouch® Plus system (FT)
  Interventions: Device: Advanced Pneumatic Compression Device (APCD)
- Usual Care (Active Comparator): Complete Decongestive Therapy (CDT) directed by a lymphedema therapist and any additional adjunctive measures as prescribed by the lymphedema therapist
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Advanced Pneumatic Compression Device (APCD) — Once daily treatment with Flexitouch Plus.
  Other Names: Flexitouch; Flexitouch Plus
  Arms: Advanced Pneumatic Compression Device (APCD)
Other: Usual Care — Usual care consists of a two-phase CDT. Phase 1 includes consultation with a lymphedema therapist, patient education, MLD, compression garments or bandages, skin care techniques, and a program of exercises and postural recommendations. Phase 2 consists of ongoing self-care, where patients conduct a life-long program of disease management that mimics the program in phase 1.
  Other Names: Complete Decongestive Therapy (CDT); Manual Lymphatic Drainage (MLD)
  Arms: Usual Care

SUMMARY:
To compare the effectiveness of an APCD to Usual Care in the management of lymphedema and fibrosis (LEF) in head and neck cancer (HNC) survivors.

DETAILED DESCRIPTION:
Aim 1:

To compare the short-term and long-term effectiveness of self-administered APCD therapy versus Usual Care in HNC survivors with treatment naive LEF on anatomical measures of internal and external LEF. Baseline measures will be obtained at the start of therapy. Short-term effectiveness will be evaluated at 2 months and long-term effectiveness will be evaluated at 4 and 6 months. Hypothesis: the APCD therapy will be associated with greater short-term and long-term reduction in anatomical measures of LEF.

Aim 2:

To compare the short-term and long-term effectiveness of self-administered APCD therapy versus Usual Care in HNC survivors with treatment naive LEF on patient reported biopsychosocial outcome measures impacted by LEF. Outcome measures will include: 1) symptom burden, 2) symptom burden and functional impairment, 3) quality of life (QOL), 4) work and activity, 5) perceived self-management capacity, 6) body image, and 7) diet modifications. Baseline measures will be obtained at the start of therapy. Short-term effectiveness will be evaluated at 2 months and long-term effectiveness will be evaluated at 4 and 6 months. Hypothesis: the APCD therapy will be associated with greater short-term and long-term improvement in patient reported biopsychosocial outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Pathologically confirmed cancer of the HNC (larynx, pharynx, oral cavity, paranasal sinuses, major salivary glands, and HNC of unknown primary)
3. Completed curative intent cancer therapy with no evidence of active cancer at time of study enrollment
4. A diagnosis of either internal or external head and neck lymphedema
5. At least one core lymphedema associated symptom of ≥ 4 out of 10 at the time of study screening
6. Must be able and willing to participate in all aspects of the study and provide informed consent prior to study participation
7. Must be able to speak and understand English

Exclusion Criteria:

1. Previous APCD or Usual Care treatment for HNC LEF
2. Acute facial infection (e.g., facial or parotid gland abscess)
3. Known carotid sinus hypersensitivity syndrome
4. Symptomatic carotid artery disease, as manifested by a recent transient ischemic attack (within 30 days), ischemic stroke, or amaurosis fugax (monocular visual ischemic symptoms or blindness)
5. Internal jugular venous thrombosis (within 3 months)
6. Patient is pregnant or trying to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Reduction in Swelling/Inflammation - Endoscopy | Changes between Baseline, 2 months, 4 months, 6 months
  The change in percent of sites with visible swelling and inflammation as assessed via endoscopy (using Modified Patterson Scale). The range for each anatomical structure includes 1-4: Normal, Mild, Moderate, and Severe. A lower score means a better outcome. A greater negative value indicates a greater reduction in swelling. Total score range: 0-100%
Reduction in Swelling/Imaging - CT | Changes between Baseline, 2 months, 6 months
  The changes in fat stranding, epiglottic thickness, and prevertebral soft tissue (PVST) using the CT Lymphedema and Fibrosis Assessment Tool (CT-LEFAT). The range for fat stranding includes 0-2: Normal, Mild Changes, Advanced Changes. A lower score means a better outcome. Epiglottis and PVST are measured in mm. A lower measurement means a better outcome.
Reduction in Swelling/Inflammation - Grading of External Lymphedema | Changes between Baseline, 2 months, 4 months, 6 months
  The presence of swelling and inflammation as assessed through grading of external lymphedema via the Head and Neck Lymphedema and Fibrosis Assessment criteria (HNLEF). A total of 9 sites are evaluated for the presence of lymphedema and graded from 1 (mild) to 3 (severe) at each site. The number of sites ranged from 0-9 with a total severity score ranging from 0-27. A lower score indicates a better outcome. A greater negative value indicates a greater reduction in swelling.
Reduction in Swelling/Inflammation - Digital Photography | Changes between Baseline, 2 months, 4 months, 6 months
  The presence of swelling and inflammation are assessed by digital photography. A lower value means a better outcome. A greater negative value indicates a greater reduction in swelling. Three views are scored each with 30 grids. The percentage of views with visible swelling was determined. The score ranges from 0-100%.
Symptom Burden - Lymphedema Symptom Intensity and Distress Survey | Changes between Baseline, 2 months, 4 months, 6 months
  Lymphedema Symptom Intensity and Distress Survey-Head and Neck (LSIDS-HN) assesses the measurement characteristics of a symptom burden for participants with head and neck lymphedema. Each symptom is rated on intensity and distress using a 5-point scale. A maximum response for any symptom within a given cluster will be used for the analysis. The total score ranged from 0-10. The values represent a change from baseline. A lower score means a better outcome.
Symptom Burden and Functional Impairment - Vanderbilt Head and Neck Symptom Survey | Changes between Baseline, 2 months, 4 months, 6 months
  Vanderbilt Head and Neck Symptom Survey plus General Symptom Survey (VHNSS plus GSS) assesses symptom burden and functional impairment. Values represent a median score change from baseline. Score range: 0-10. A lower score indicates a better outcome. A more negative value indicates a greater change from baseline.
Quality of Life - Linear Analog Self-Assessment | Changes between Baseline, 2 months, 4 months, 6 months
  Quality of life is assessed using the Linear Analog Self-Assessment. The total score for the assessment ranges from 0-50. Each category represents a change in score from the baseline visit which ranged from positive 4 to negative 4. A positive change indicates an improvement.
Work and Activity - Work Productivity and Activity Impairment Questionnaire | Changes between Baseline, 2 months, 4 months, 6 months
  Work Productivity and Activity Impairment Questionnaire (WPAIQ) PRO assessment asks questions about work and activity impairment due to lymphedema and other health problems. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes. Total score range: 0-100%
Perceived self-management capacity - Perceived Medical Condition Self-Management Scale (PMCSMS) | Changes between Baseline, 2 months, 4 months, 6 months
  The 8-item Perceived Medical Condition Self-Management Scale (PMCSMS) is intended to measure patients' belief that they are capable of carrying out the self-management behaviors required by their medical condition. The scale is composed of four positively worded items and four negatively worded items, each rated on a five-point Likert scale (1=Strongly Disagree to 5=Strongly Agree). Negatively worded items are reversed scored, yielding a total score ranging from 8 to 40, with a higher score indicating stronger belief of perceived self-management competence.
Body image - Body Image Quality of Life Inventory (BIQLI) | Changes between Baseline, 2 months, 4 months, 6 months
  Body Image Quality Life Inventory (BIQLI) assesses participants' body image using 7 point scale ranging from -3 (very negative) to +3 (very positive). Score range: -57 to 57. A higher score indicates a better outcome.
Diet modifications - Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24) | Changes between Baseline, 2 months, 4 months, 6 months
  Diet modifications will be assessed using the Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24). The ASA24 is a tool from National Cancer Institute (NCI) that enables multiple automatically coded self-administered 24-hour recalls and food records. Changes in total caloric intake, fat, carbohydrate, fiber, sugars, and protein will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Principal Investigator — Vanderbilt University Medical Center; Sheila Ridner, RN, PhD, Principal Investigator — Vanderbilt University
Locations (10):
- United States (10):
  - University of Alabama, Birmingham, Alabama
  - Rush University Medical Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Richmond University Medical Center, Staten Island, New York
  - Montefiore Medical Center, The Bronx, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Advanced Head & Neck Rehabilitation Center of Texas, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murphy BA, Smith DK, Kline-Quiroz CM, Jensen KM, Sukari AW, Bhayani MK, Mehta V, Quon H, Shah JL, Willey CD, Dunlap NE, Lee HK, Aulino JM, Ridner SH. Short-Term Outcomes of Advanced Pneumatic Compression Device Versus Usual Care Therapy for Head and Neck Cancer-Related Lymphedema: A Multi-Site Randomized Clinical Trial. Head Neck. 2026 Jan 23. doi: 10.1002/hed.70155. Online ahead of print. PMID 41574713